CLINICAL TRIAL: NCT00005271
Title: INTERMAP: International Population Study on Macronutrients and BP
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1155; R01HL050490 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — 24 hour urine collection among all participants
Oversight: Data Monitoring Committee: No

SUMMARY:
To investigate the relationship between dietary factors, especially macronutrients, and blood pressure in an international, multicenter observational study. A particular focus is to help elucidate the role of these dietary factors in accounting for the even more adverse blood pressure patterns of less educated population strata, especially in the United States, in both less educated Blacks and whites.

DETAILED DESCRIPTION:
BACKGROUND:

Overall study findings are to be used to estimate favorable impact on blood pressure of multiple improvements in nutrition by populations. The investigators state that this should aid in making additional dietary recommendations toward the goal of primary prevention of hypertension and shifting blood pressure distributions downward to avoid excess risk associated with present levels generally above optimal.

DESIGN NARRATIVE:

INTERMAP's cross-sectional design is patterned after the tested INTERSALT model: a large sample size of 4,680 persons, half men and half women, ages 40-59 from 17 population samples of varied ethnicity, socioeconomic status (SES) and dietary habits in four countries (China, Japan, United Kingdom and the United States). There were eight United States INTERMAP centers. Specific aims involve elucidating influences on blood pressure of the amount and type of protein, lipids, carbohydrates, and also amino acids, calcium, magnesium, antioxidants, fiber, and caffeine. Primary hypotheses tested, with control for body mass index (BMI), intake of alcohol, age, sex, and other confounders are as follow: dietary protein is inversely related to blood pressure; inverse relations between education and blood pressure are significantly accounted for by education-related differences in dietary protein intake; there is a direct relation to blood pressure of dietary saturated fatty acids, cholesterol, Keys score, starch; there is an inverse relation of polyunsaturated fatty acids and polyunsaturated/saturated fatty acids. Randomly selected participants provide one timed 24-hr. urine collection for assessment of sodium, potassium, creatine, and urea, and complete four 24-hr. dietary recalls. Blood pressure was measured eight times at each of four clinic visits, with standardization and strict quality control of all procedures.

The study is coordinated by two Coordinating Centers--Northwestern University, Chicago and London School of Hygiene & Tropical Medicine. Urinary determinations are made at a Central Laboratory in Leuven, Belgium. Twenty-four hour dietary recalls are converted into nutrients with use of the Nutrition Data System of the University of Minnesota's Nutrition Coordinating Center. Data analyses to test hypotheses are done at the London Coordinating Center.

Recruitment and data collection began in July, 1996 through January, 1997. The main statistical analytic method is multivariate regression analysis. The study was renewed in FY 2000 and in FY 2004 to continue analysis of the data through August, 2009.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals
* Men and women
* Age 40-59 years
* Willing to collect 24 hour urine and return to clinic for second follow-up visit

Exclusion Criteria:

* Existing disease
* Unwilling to provide 24 hour urine collections
* Unable to attend follow-up visits
* Unable to recall dietary intake

Ages: 40 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The INTERMAP study population includes 4,680 men and women ages 40-59 who were recruited from 17 population samples of diverse ethnicity/ SES/ eating practices in four countries (China, Japan, UK, USA).
Sampling Method: Probability Sample
Enrollment: 4680 (Actual)
Dates: Start 1995-07; Primary Completion 2009-08 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Blood pressure measurement relative to diet. | 15 years
  Ongoing comparisons of different nutrients, urinary sodium and blood pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Appel, Principal Investigator — Johns Hopkins University; Daniel Jones, Principal Investigator — University of Mississippi Medical Center; Darwin Labarthe, Principal Investigator — University of Texas; Beatriz Rodriguez, Principal Investigator — University of Hawaii at Manoa; Jeremiah Stamler, Principal Investigator — Northwestern University; Linda Van Horn, Principal Investigator — Northwestern University

REFERENCES:
- [Background] Stamler J, Elliott P, Dennis B, Dyer AR, Kesteloot H, Liu K, Ueshima H, Zhou BF; INTERMAP Research Group. INTERMAP: background, aims, design, methods, and descriptive statistics (nondietary). J Hum Hypertens. 2003 Sep;17(9):591-608. doi: 10.1038/sj.jhh.1001603. PMID 13679950
- [Background] Beevers DG, Stamler J. Background to the INTERMAP study of nutrients and blood pressure. J Hum Hypertens. 2003 Sep;17(9):589-90. doi: 10.1038/sj.jhh.1001609. No abstract available. PMID 13679949
- [Background] Dennis B, Stamler J, Buzzard M, Conway R, Elliott P, Moag-Stahlberg A, Okayama A, Okuda N, Robertson C, Robinson F, Schakel S, Stevens M, Van Heel N, Zhao L, Zhou BF; INTERMAP Research Group. INTERMAP: the dietary data--process and quality control. J Hum Hypertens. 2003 Sep;17(9):609-22. doi: 10.1038/sj.jhh.1001604. PMID 13679951
- [Background] Zhou BF, Stamler J, Dennis B, Moag-Stahlberg A, Okuda N, Robertson C, Zhao L, Chan Q, Elliott P; INTERMAP Research Group. Nutrient intakes of middle-aged men and women in China, Japan, United Kingdom, and United States in the late 1990s: the INTERMAP study. J Hum Hypertens. 2003 Sep;17(9):623-30. doi: 10.1038/sj.jhh.1001605. PMID 13679952
- [Background] Dyer AR, Elliott P, Stamler J, Chan Q, Ueshima H, Zhou BF; INTERMAP Research Group. Dietary intake in male and female smokers, ex-smokers, and never smokers: the INTERMAP study. J Hum Hypertens. 2003 Sep;17(9):641-54. doi: 10.1038/sj.jhh.1001607. PMID 13679954
- [Background] Stamler J, Elliott P, Appel L, Chan Q, Buzzard M, Dennis B, Dyer AR, Elmer P, Greenland P, Jones D, Kesteloot H, Kuller L, Labarthe D, Liu K, Moag-Stahlberg A, Nichaman M, Okayama A, Okuda N, Robertson C, Rodriguez B, Stevens M, Ueshima H, Horn LV, Zhou B. Higher blood pressure in middle-aged American adults with less education-role of multiple dietary factors: the INTERMAP study. J Hum Hypertens. 2003 Sep;17(9):655-775. doi: 10.1038/sj.jhh.1001608. PMID 13679955
- [Background] Conway R, Robertson C, Dennis B, Stamler J, Elliott P; INTERMAP Research Group. Standardised coding of diet records: experiences from INTERMAP UK. Br J Nutr. 2004 May;91(5):765-71. doi: 10.1079/BJN20041095. PMID 15152639
- [Background] Zhao L, Stamler J, Yan LL, Zhou B, Wu Y, Liu K, Daviglus ML, Dennis BH, Elliott P, Ueshima H, Yang J, Zhu L, Guo D; INTERMAP Research Group. Blood pressure differences between northern and southern Chinese: role of dietary factors: the International Study on Macronutrients and Blood Pressure. Hypertension. 2004 Jun;43(6):1332-7. doi: 10.1161/01.HYP.0000128243.06502.bc. Epub 2004 Apr 26. PMID 15117915
- [Background] Dyer AR, Greenland P, Elliott P, Daviglus ML, Claeys G, Kesteloot H, Chan Q, Ueshima H, Stamler J; INTERMAP Research Group. Estimating laboratory precision of urinary albumin excretion and other urinary measures in the International Study on Macronutrients and Blood Pressure. Am J Epidemiol. 2004 Aug 1;160(3):287-94. doi: 10.1093/aje/kwh196. PMID 15258002
- [Background] Dyer AR, Greenland P, Elliott P, Daviglus ML, Claeys G, Kesteloot H, Ueshima H, Stamler J; INTERMAP Research Group. Evaluation of measures of urinary albumin excretion in epidemiologic studies. Am J Epidemiol. 2004 Dec 1;160(11):1122-31. doi: 10.1093/aje/kwh326. PMID 15561992
- [Background] Daviglus ML, Greenland P, Stamler J, Elliott P, Appel LJ, Carnethon MR, Chan Q, Claeys G, Kesteloot H, Miura K, Nakagawa H, Pirzada A, Steffen L, Yan LL, Zhou B, Dyer AR. Relation of nutrient intake to microalbuminuria in nondiabetic middle-aged men and women: International Population Study on Macronutrients and Blood Pressure (INTERMAP). Am J Kidney Dis. 2005 Feb;45(2):256-66. doi: 10.1053/j.ajkd.2004.11.005. PMID 15685502
- [Background] Elliott P, Stamler J, Dyer AR, Appel L, Dennis B, Kesteloot H, Ueshima H, Okayama A, Chan Q, Garside DB, Zhou B. Association between protein intake and blood pressure: the INTERMAP Study. Arch Intern Med. 2006 Jan 9;166(1):79-87. doi: 10.1001/archinte.166.1.79. PMID 16401814
- [Derived] Oude Griep LM, Chekmeneva E, Van Horn L, Chan Q, Daviglus ML, Frost G, Holmes E, Ebbels TM, Elliott P. A Metabolome Wide Association Study of Fruit and Vegetable Consumption and Associations with Cardiovascular Disease Risk Factors: The International Study of Macro-/Micronutrients and Blood Pressure (INTERMAP) Study. J Nutr. 2025 Jan;155(1):122-131. doi: 10.1016/j.tjnut.2024.11.004. Epub 2024 Nov 12. PMID 39536968
- [Derived] Gibson R, Aljuraiban GS, Oude Griep LM, Vu TH, Steffen LM, Appel LJ, Rodriguez BL, Daviglus ML, Elliott P, Van Horn L, Chan Q. Relationship of calcium and magnesium intakes with the dietary approaches to stop hypertension score and blood pressure: the International Study of Macro/micronutrients and Blood Pressure. J Hypertens. 2024 May 1;42(5):789-800. doi: 10.1097/HJH.0000000000003648. Epub 2023 Dec 20. PMID 38164982
- [Derived] Salman E, Kadota A, Okami Y, Kondo K, Yoshita K, Okuda N, Nakagawa H, Saitoh S, Sakata K, Okayama A, Chan Q, Elliott P, Stamler J, Ueshima H, Miura K; INTERMAP Research Group. Investigation of the urinary sodium-to-potassium ratio target level based on the recommended dietary intake goals for the Japanese population: The INTERMAP Japan. Hypertens Res. 2022 Dec;45(12):1850-1860. doi: 10.1038/s41440-022-01007-x. Epub 2022 Nov 8. PMID 36344663
- [Derived] Chan Q, Wren GM, Lau CE, Ebbels TMD, Gibson R, Loo RL, Aljuraiban GS, Posma JM, Dyer AR, Steffen LM, Rodriguez BL, Appel LJ, Daviglus ML, Elliott P, Stamler J, Holmes E, Van Horn L. Blood pressure interactions with the DASH dietary pattern, sodium, and potassium: The International Study of Macro-/Micronutrients and Blood Pressure (INTERMAP). Am J Clin Nutr. 2022 Jul 6;116(1):216-229. doi: 10.1093/ajcn/nqac067. PMID 35285859
- [Derived] Aljuraiban G, Chan Q, Gibson R, Stamler J, Daviglus ML, Dyer AR, Miura K, Wu Y, Ueshima H, Zhao L, Van Horn L, Elliott P, Oude Griep LM; INTERMAP Research Group. Association between plant-based diets and blood pressure in the INTERMAP study. BMJ Nutr Prev Health. 2020 Jul 8;3(2):133-142. doi: 10.1136/bmjnph-2020-000077. eCollection 2020 Dec. PMID 33521522
- [Derived] Gibson R, Lau CE, Loo RL, Ebbels TMD, Chekmeneva E, Dyer AR, Miura K, Ueshima H, Zhao L, Daviglus ML, Stamler J, Van Horn L, Elliott P, Holmes E, Chan Q. The association of fish consumption and its urinary metabolites with cardiovascular risk factors: the International Study of Macro-/Micronutrients and Blood Pressure (INTERMAP). Am J Clin Nutr. 2020 Feb 1;111(2):280-290. doi: 10.1093/ajcn/nqz293. PMID 31782492
- [Derived] Zhou L, Stamler J, Chan Q, Van Horn L, Daviglus ML, Dyer AR, Miura K, Okuda N, Wu Y, Ueshima H, Elliott P, Zhao L; INTERMAP Research Group. Salt intake and prevalence of overweight/obesity in Japan, China, the United Kingdom, and the United States: the INTERMAP Study. Am J Clin Nutr. 2019 Jul 1;110(1):34-40. doi: 10.1093/ajcn/nqz067. PMID 31111867
- [Derived] Wen X, Zhou L, Stamler J, Chan Q, Van Horn L, Daviglus ML, Dyer AR, Elliott P, Ueshima H, Miura K, Okuda N, Wu Y, Zhao L. Agreement between 24-h dietary recalls and 24-h urine collections for estimating sodium intake in China, Japan, UK, USA: the International Study of Macro- and Micro-nutrients and Blood Pressure. J Hypertens. 2019 Apr;37(4):814-819. doi: 10.1097/HJH.0000000000001941. PMID 30817463
- [Derived] Stamler J, Chan Q, Daviglus ML, Dyer AR, Van Horn L, Garside DB, Miura K, Wu Y, Ueshima H, Zhao L, Elliott P; INTERMAP Research Group. Relation of Dietary Sodium (Salt) to Blood Pressure and Its Possible Modulation by Other Dietary Factors: The INTERMAP Study. Hypertension. 2018 Apr;71(4):631-637. doi: 10.1161/HYPERTENSIONAHA.117.09928. PMID 29507099
- [Derived] Aljuraiban GS, Chan Q, Oude Griep LM, Brown IJ, Daviglus ML, Stamler J, Van Horn L, Elliott P, Frost GS; INTERMAP Research Group. The impact of eating frequency and time of intake on nutrient quality and Body Mass Index: the INTERMAP Study, a Population-Based Study. J Acad Nutr Diet. 2015 Apr;115(4):528-36.e1. doi: 10.1016/j.jand.2014.11.017. Epub 2015 Jan 22. PMID 25620753
- [Derived] Chan Q, Stamler J, Brown IJ, Daviglus ML, Van Horn L, Dyer AR, Oude Griep LM, Miura K, Ueshima H, Zhao L, Nicholson JK, Holmes E, Elliott P; INTERMAP Research Group. Relation of raw and cooked vegetable consumption to blood pressure: the INTERMAP Study. J Hum Hypertens. 2014 Jun;28(6):353-9. doi: 10.1038/jhh.2013.115. Epub 2013 Nov 21. PMID 24257514
- [Derived] Stamler J, Brown IJ, Yap IK, Chan Q, Wijeyesekera A, Garcia-Perez I, Chadeau-Hyam M, Ebbels TM, De Iorio M, Posma J, Daviglus ML, Carnethon M, Holmes E, Nicholson JK, Elliott P; INTERMAP Research Group. Dietary and urinary metabonomic factors possibly accounting for higher blood pressure of black compared with white Americans: results of International Collaborative Study on macro-/micronutrients and blood pressure. Hypertension. 2013 Dec;62(6):1074-80. doi: 10.1161/HYPERTENSIONAHA.113.01810. Epub 2013 Oct 7. PMID 24101663
- [Derived] Oude Griep LM, Stamler J, Chan Q, Van Horn L, Steffen LM, Miura K, Ueshima H, Okuda N, Zhao L, Daviglus ML, Elliott P; INTERMAP Research Group. Association of raw fruit and fruit juice consumption with blood pressure: the INTERMAP Study. Am J Clin Nutr. 2013 May;97(5):1083-91. doi: 10.3945/ajcn.112.046300. Epub 2013 Apr 3. PMID 23553162